CLINICAL TRIAL: NCT04565795
Title: URIPRENE: Clinical Study to Evaluate the Safety and Device Performance of the ADVA-Tec Uriprene® Degradable Temporary Ureteral Stent Following Uncomplicated Ureteroscopy
Brief Title: Safety and Device Performance of the Uriprene® Degradable Temporary Ureteral Stent Following Uncomplicated Ureteroscopy
Acronym: URIPRENE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adva-Tec (Industry)
Collaborators: Northwest Clinical Research Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0001
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Ureteral Diseases
Keywords: ureteral stent
MeSH Terms: conditions — Ureteral Diseases

STUDY DESIGN:
Intervention Model Description: Patients with clinical symptoms consistent with unilateral ureteral or renal stone fragments post-uncomplicated ureteroscopy (UURS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Placement of ureteral stent post ureteroscopy (Experimental): Subjects with unilateral ureteral or renal stone fragments who have undergone an uncomplicated ureteroscopy (UURS)
  Interventions: Device: Uriprene® Degradable Temporary Ureteral Stent

INTERVENTIONS:
Device: Uriprene® Degradable Temporary Ureteral Stent — Assess adequate intervention-free drainage during use and the time to complete degradation or the passage of stent fragments/segments from the urinary system by radiological assessment.

SUMMARY:
A prospective, multi-center, non-randomized trial to demonstrate safety and device performance of the ADVA-Tec Uriprene® Degradable Temporary Ureteral Stent.

DETAILED DESCRIPTION:
A prospective, multi-center, non-randomized trial to demonstrate safety and device performance of the ADVA-Tec Uriprene® Degradable Temporary Ureteral Stent. The study is intended to assess the safety and efficacy of the Uriprene® Stent by assessing adequate intervention-free drainage during use and the time to complete degradation or the passage of stent fragments/segments from the urinary system by radiological assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are >21, <80 years of age; inclusive of males and females.
2. Subjects with unilateral ureteral or renal stones who have undergone a successful, uncomplicated ureteroscopy (UURS).
3. Subjects with asymptomatic, contralateral renal stones in sizes <4mm WHICH ARE NOT IN THE RENAL PELVIS OR URETER and who have had uncomplicated ureteroscopy (UURS) can be included. If, during the course of treatment of the target ureter with the Uriprene stent the patient's asymptomatic stone becomes symptomatic and requires treatment, the patient can only be managed with standard of care treatment including the use of an approved ureteral stent, if necessary.
4. Subjects with a height and body size able to accommodate a 20, 22, 24, 26, 28, or 30 mm long ureteral stent, as judged by the Investigator.
5. Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and are willing to undergo all follow-up assessments according to the specified schedule.

Exclusion Criteria:

1. Subjects with a history of an anatomical abnormality of the urinary tract.
2. Presence of ureteral fistula.
3. Presence of urothelial cancer, ureteral tumor, or renal tumor.
4. Presence of extrinsic compression of the ureter.
5. Presence of ureteral blockage or stricture.
6. Bladder outlet obstruction or neurogenic bladder.
7. Subjects with known/diagnosed overactive bladder (OAB).
8. Subjects with known/diagnosed urge urinary incontinence (UUI).
9. Subjects with a known, active upper or lower urinary tract infection at the time of stent insertion.
10. Subjects with creatinine level of ˃2.5 mg/dl.
11. Pregnant or lactating women, or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
12. Impacted ureteral stones still in place and/or incomplete stone fragmentation.
13. Ureteral perforation.
14. Staghorn calculi.
15. Subjects with a solitary kidney.
16. History of bleeding diathesis or currently taking blood thinners such as warfarin (anti- platelet agents are allowed).
17. Contrast allergy that cannot be adequately pre-treated.
18. Subject has known severe psychiatric disorder, substance abuse, or other reason for being unable to follow trial follow-up instructions or unable to reliably complete patient questionnaires.
19. Any condition, in the opinion of the investigator, that would deem a subject as ineligible for treatment with the Uriprene® Stent.
20. Subject has a known significant concomitant illness with a life expectancy of <1 year.
21. Subject is known to be currently enrolled in another investigational trial.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint defined as the presence of the stent during the first 48 hours | 48 hours
  Study Success defined as adequate short-term urine drainage, defined as the presence of the stent in the ureter and the lack of surgical or invasive intervention to treat symptoms in the stented ureter during the first 48 hours following placement.
Primary Safety Endpoint defined as assessment of adverse events through 90 days | 90 days
  Assessment of Adverse Events through the 90-day follow-up period (incidence, relationship to device and severity) compared to the historical control degradable ureteral stent and plastic ureteral stents

SECONDARY OUTCOMES:
Overall Clinical Success | 90 days
  Adequate urine drainage with no intervention and no definitely device-related serious adverse events (SAEs) throughout the 90-day follow-up period.
Technical success of the device | 90 days
  Complete degradation/elimination of the stent from the urinary system within 90 days as measured by radiological assessment.
Tolerability of device presence defined as assessment of pain via the Ureteral Stent Symptom Questionnaire (USSQ) and Patient Diary for pain medications. | 90 days
  Tolerability of device presence defined as assessment of pain via the Ureteral Stent Symptom Questionnaire (USSQ) and Patient Diary for pain medications.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Humphreys, MD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No